CLINICAL TRIAL: NCT01921465
Title: Outpatient Care for Multiparas After Elective Cesarean Section: an Observational Study
Status: Completed | Type: Observational
Sponsor: Herning Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Iben Lorentzen, Midwife, Herning Hospital
Other Study IDs: 1ILorentzen; outpatientcesareanlorentzen
Record Dates: First submitted 2013-08-09; First posted 2013-08-13 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2014-02

CONDITIONS: Outpatient Care
Keywords: outpatient care; videoconferencing; elective cesarean section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- multiparas having a planned cesarean section: elective cesarean section

SUMMARY:
The purpose of the study is to evaluate whether outpatient cesarean section can be performed in multiparous women without significant decrease in the parents' sense of security .

ELIGIBILITY:
Inclusion Criteria:

* Planned elective cesarean section of multiparous women
* Singleton pregnancy
* Age of at least 18
* Gestational age between 37 and 42 weeks
* Internet access at home

Exclusion Criteria:

* Lack of consent
* Women with no or little understanding of Danish and ability to speak Danish.
* Allergies to medicine included in the pain management regimes
* Expected maternal or neonatal complications after delivery
* Birth weight of less than 2500 grams

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: multiparas having a elective cesarean section at Herning hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the parents' postnatal sense of security (PPSS) | the PPSS is measured the second week after delivery
  measured by a questionnaire sent to the parents' in the second week after delivery.

SECONDARY OUTCOMES:
ambulation time | three days
  ambulation time measured during the first three days after delivery by an accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Iben P Lorentzen, Midwife, Principal Investigator — University of Aarhus
Locations (1):
- Department of gynaecology and obstetrics, Herning Hospital, Herning, Herning, Denmark